CLINICAL TRIAL: NCT06106503
Title: Routine Chest X-ray Post Rigid Bronchoscopy for Foreign Body Extraction: is it Necessary?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Ibrahim Abdelrahman Boudy, Doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: chest xray post bronchoscopy
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Foreign Body Aspiration
MeSH Terms: conditions — Respiratory Aspiration | interventions — X-Rays; Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients will not underwent chest x-ray (Other)
  Interventions: Other: clinical examination
- patients underwent chest x-ray (Other): patients underwent chest x-ray
  Interventions: Radiation: chest x-ray

INTERVENTIONS:
Radiation: chest x-ray — chest x-ray after rigid bronchoscopy for patient with foreign body inhalation
  Arms: patients underwent chest x-ray
Other: clinical examination — no investigations well be done unless needed
  Arms: patients will not underwent chest x-ray

SUMMARY:
Airway foreign body is one of the common emergencies. Its clinical presentation is variable, ranging from a clinically asymptomatic state to dire state of respiratory failure needing urgent attention and intervention. The gold standard for management is rigid bronchoscopy (RB) under general anaesthesia. Complications that can occur during removal of foreign body include bleeding, pneumothorax and rupture of tracheobronchial tree. Complication rates are higher during foreign body removal in children. Performance of routine post bronchoscopy chest radiography (CXR) results in an extremely low diagnostic yield but nevertheless is the common clinical practice prevailing today. It has previously been suggested that routine post bronchoscopy CXR could be avoided in asymptomatic patients.

DETAILED DESCRIPTION:
* Pre-operative assessment:

  1. History taking including if there was a definite history of foreign body inhalation or not.
  2. Clinical examination including symptomatology (such as the presence or absence of choking, cyanosis, and difficulty in breathing) and Clinical signs, such as the presence or absence of air entry, crept, and rhonchi.
  3. Radiological signs, such as plain chest X-ray findings.
* operation: all patients underwent rigid bronchoscopy under general anesthesia. We used bronchoscopes of the rigid type to perform bronchoscopy. We determined the size of the bronchoscope according to the child's age. After induction of intravenous anesthesia, we performed direct laryngoscopy and inserted the bronchoscope with the help of the laryngoscope in a rotating manner and used a 0-degree telescope to locate the foreign body. Once identified, we used optical forceps to hold and to remove the foreign body. After extraction of the foreign body, we repeated bronchoscopy to check for any remaining foreign bodies as well as to examine the tracheobronchial tree for any trauma.
* Post-operative assessment:

All patients will be under observation for at least an hour after the procedure.

All patients will receive ATROVENT and PULMICORT after the procedure through a nebulizer.

All patients will be examined clinically and vital signs will be assessed be before discharge CXR will be done only if there are critical signs as cyanosis, absent or decreased air entery on one side or both or surgical emphysema Strict instructions, that if any symptoms such as cyanosis or difficulty of breathing occur, to go the nearest health care provider.

ELIGIBILITY:
Inclusion Criteria:

* All patients with strong clinical suspicion of foreign body in airway with a history of choking, cyanosis, difficulty in breathing.
* All patients with strong clinical suspicion of foreign body in airway with the presence of clinical signs, like decreased air entry, cyanosis, or crept. Patients of any age and sex who qualified for the inclusion criteria were included.

Exclusion Criteria:

* Patients underwent esophagoscope.
* Patients refused to be enrolled in research.
* Patients suffering from evident complications during the procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
chest x-ray post bronchoscopy. | 2 years
  chest x-ray post bronchoscopy is not necessary unless there are signs or symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed ayaad, professor, Study Director — Director